CLINICAL TRIAL: NCT04516499
Title: Remote Blood Biomarker Monitoring in Frontotemporal Lobar Degeneration: Neurofilament Surveillance Project (NSP)
Brief Title: Neurofilament Surveillance Project (NSP)
Status: Active, not recruiting | Type: Observational
Sponsor: The Bluefield Project to Cure Frontotemporal Dementia (Other)
Collaborators: Mayo Clinic (Other); University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: NSP001
Record Dates: First submitted 2020-08-11; First posted 2020-08-18 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Frontotemporal Dementia; Frontotemporal Lobar Degeneration; FTD-GRN; FTD; FTLD
Keywords: C9orf72; GRN; MAPT
MeSH Terms: conditions — Frontotemporal Dementia; Frontotemporal Lobar Degeneration; Frontotemporal Dementia With Motor Neuron Disease

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma will be extracted from participant's whole blood. The plasma will be analyzed for the levels of neurofilament light chain and other potential biomarkers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- f-FTLD mutation carriers: All participants must be from a family with f-FTLD mutations. The f-FTLD mutation carrier group members will have their genetic status tested and included in this group if a f-FTLD mutation is observed. Participants do not need to know or be told their genetic status.
- Non-mutation carriers from families with f-FTLD mutations: All participants must be from a family with f-FTLD mutations. The non-mutation carrier group members will have their genetic status tested and included in this group if they do not have a f-FTLD mutation. Participants do not need to know or be told their genetic status.

SUMMARY:
This is a biomarker study designed to collect and analyze blood specimens from individuals carrying known familial frontotemporal lobar degeneration (f-FTLD) mutations compared to a control group of individuals without known f-FTLD mutations. The NSP is an ancillary study to the ARTFL LEFFTDS Longitudinal Frontotemporal Lobar Degeneration" (ALLFTD) study, NCT04363684. More information can be found at https://www.allftd.org/.

DETAILED DESCRIPTION:
Frontotemporal Lobar Degeneration (FTLD), a group of clinically heterogeneous neurodegenerative diseases characterized by progressive deterioration of the frontal and temporal cortices as well as basal ganglia and brainstem structures, is a common cause of neurodegenerative dementia in people who are less than 60 years old at onset. It is uniformly fatal. FTLD is a rare disease, with an estimated prevalence of approximately 5-22 per 100,000. There are no approved treatments, however several investigational agents are in human trials and a variety of novel agents are poised to enter human development. Experience from other neurodegenerative diseases suggests that potential disease modifying treatments are most likely to be efficacious if initiated before the onset of symptoms.

Approximately 25% of FTLD cases are familial (f-FTLD) and due to autosomal dominant mutations in one of three genes: C9orf72, progranulin (GRN) or microtubule associated protein tau (MAPT). Many of the new therapies entering the clinic directly target one of these genetic causes and raise the possibility that the clinical features of FTLD could be delayed or prevented in these individuals if an efficacious therapy was initiated prior to the onset of symptoms. The major barrier to determining efficacy of novel therapeutic agents for f-FTLD in such prevention trials is the lack of an endpoint that can indicate therapeutic efficacy prior to the onset of symptoms. Our preliminary data strongly suggest that plasma neurofilament light chain (NfL) could serve as such a biomarker.

This non-interventional study is in preparation for pivotal clinical trials. Up to 335 participants will provide blood remotely via visits from traveling mobile research nurses four times a year for three years (4355 samples total) to enable the observation of peripheral NfL levels longitudinally during disease onset and progression, with the ultimate goal of qualifying plasma NfL as an endpoint for f-FTLD prevention trials. The NSP study is an ancillary study to ALLFTD, and biomarker data collected in the NSP will be correlated with ALLFTD clinical data. More information on the NSP study may be found at https://www.allftd.org/nsp.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female
2. Ages 18-85
3. Provision of signed and dated informed consent form
4. Stated willingness to comply with all study procedures and availability for the duration of the study
5. Is enrolled in the longitudinal arm of ALLFTD
6. Is a member of a family with a known mutation in C9orf72, GRN or MAPT

Exclusion Criteria:

1. Any permanent contra-indication to repeated blood draws, such as poor venous access.
2. Any conditions or circumstances which, in the opinion of the investigator, would not allow participation in the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study is an ancillary study to ALLFTD. Thus, all NSP participants will be recruited directly from the longitudinal arm of ALLFTD.
  Roughly equivalent numbers of participants will be enrolled from each of the following groups:
  * Members of families with known mutations in C9orf72
  * Members of families with known mutations in GRN
  * Members of families with known mutations in MAPT
  Although participant must be from a family with a known mutation, the participant themselves need not know their personal mutation status.
Sampling Method: Non-Probability Sample
Enrollment: 342 (Actual)
Dates: Start 2020-09-02 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Neurofilament Light Chain Levels | 36 months
  To determine the longitudinal stability of plasma neurofilament light chain (NfL) measured every 3 months for 36 months in individuals at-risk for symptomatic FTLD

SECONDARY OUTCOMES:
Intersubject variability of plasma NfL measurements | 36 months
  Concentration of plasma neurofilament light chain protein
Logistics measure | 36 months
  Participant compliance with scheduled remote blood collection and sample processing

OTHER OUTCOMES:
Clinical and MRI correlates | 36 months
  To evaluate ALLFTD collected clinical and magnetic resonance imaging (MRI) neuroimaging correlates with plasma NfL levels in asymptomatic and symptomatic f-FTLD mutation carriers
Other biomarker evaluation | 36 months
  To measure other novel blood biomarkers of neurodegeneration yet to be determined

CONTACTS AND LOCATIONS:
Overall Officials: Adam Boxer, MD, PhD, Principal Investigator — University of California, San Francisco; Bradley Boeve, MD, Principal Investigator — Mayo Clinic; Howie Rosen, MD, Principal Investigator — University of California, San Francisco; Laura Mitic, PhD, Study Director — The Bluefield Project to Cure Frontotemporal Dementia
Locations (8):
- United States (8):
  - University of California, San Francisco, San Francisco, California
  - Mayo Clinic Florida, Jacksonville, Florida
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Massachusetts General Hospital, Charlestown, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Washington University in St. Louis, St Louis, Missouri
  - Columbia University, New York, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided
Please consult with ALLFTD regarding individual participant data.

REFERENCES:
- [Background] Saracino D, Dorgham K, Camuzat A, Rinaldi D, Rametti-Lacroux A, Houot M, Clot F, Martin-Hardy P, Jornea L, Azuar C, Migliaccio R, Pasquier F, Couratier P, Auriacombe S, Sauvee M, Boutoleau-Bretonniere C, Pariente J, Didic M, Hannequin D, Wallon D; French Research Network on FTD/FTD-ALS; PREV-DEMALS and Predict-PGRN study groups; Colliot O, Dubois B, Brice A, Levy R, Forlani S, Le Ber I. Plasma NfL levels and longitudinal change rates in C9orf72 and GRN-associated diseases: from tailored references to clinical applications. J Neurol Neurosurg Psychiatry. 2021 Dec;92(12):1278-1288. doi: 10.1136/jnnp-2021-326914. Epub 2021 Aug 4. PMID 34349004
- [Background] Wilke C, Reich S, van Swieten JC, Borroni B, Sanchez-Valle R, Moreno F, Laforce R, Graff C, Galimberti D, Rowe JB, Masellis M, Tartaglia MC, Finger E, Vandenberghe R, de Mendonca A, Tagliavini F, Santana I, Ducharme S, Butler CR, Gerhard A, Levin J, Danek A, Otto M, Frisoni G, Ghidoni R, Sorbi S, Bocchetta M, Todd E, Kuhle J, Barro C; Genetic Frontotemporal dementia Initiative (GENFI); Rohrer JD, Synofzik M. Stratifying the Presymptomatic Phase of Genetic Frontotemporal Dementia by Serum NfL and pNfH: A Longitudinal Multicentre Study. Ann Neurol. 2022 Jan;91(1):33-47. doi: 10.1002/ana.26265. Epub 2021 Nov 29. PMID 34743360
- [Background] Rojas JC, Wang P, Staffaroni AM, Heller C, Cobigo Y, Wolf A, Goh SM, Ljubenkov PA, Heuer HW, Fong JC, Taylor JB, Veras E, Song L, Jeromin A, Hanlon D, Yu L, Khinikar A, Sivasankaran R, Kieloch A, Valentin MA, Karydas AM, Mitic LL, Pearlman R, Kornak J, Kramer JH, Miller BL, Kantarci K, Knopman DS, Graff-Radford N, Petrucelli L, Rademakers R, Irwin DJ, Grossman M, Ramos EM, Coppola G, Mendez MF, Bordelon Y, Dickerson BC, Ghoshal N, Huey ED, Mackenzie IR, Appleby BS, Domoto-Reilly K, Hsiung GR, Toga AW, Weintraub S, Kaufer DI, Kerwin D, Litvan I, Onyike CU, Pantelyat A, Roberson ED, Tartaglia MC, Foroud T, Chen W, Czerkowicz J, Graham DL, van Swieten JC, Borroni B, Sanchez-Valle R, Moreno F, Laforce R, Graff C, Synofzik M, Galimberti D, Rowe JB, Masellis M, Finger E, Vandenberghe R, de Mendonca A, Tagliavini F, Santana I, Ducharme S, Butler CR, Gerhard A, Levin J, Danek A, Otto M, Sorbi S, Cash DM, Convery RS, Bocchetta M, Foiani M, Greaves CV, Peakman G, Russell L, Swift I, Todd E, Rohrer JD, Boeve BF, Rosen HJ, Boxer AL; ALLFTD and GENFI consortia. Plasma Neurofilament Light for Prediction of Disease Progression in Familial Frontotemporal Lobar Degeneration. Neurology. 2021 May 4;96(18):e2296-e2312. doi: 10.1212/WNL.0000000000011848. Epub 2021 Apr 7. PMID 33827960
- [Background] Gendron TF, Heckman MG, White LJ, Veire AM, Pedraza O, Burch AR, Bozoki AC, Dickerson BC, Domoto-Reilly K, Foroud T, Forsberg LK, Galasko DR, Ghoshal N, Graff-Radford NR, Grossman M, Heuer HW, Huey ED, Hsiung GR, Irwin DJ, Kaufer DI, Leger GC, Litvan I, Masdeu JC, Mendez MF, Onyike CU, Pascual B, Ritter A, Roberson ED, Rojas JC, Tartaglia MC, Wszolek ZK, Rosen H, Boeve BF, Boxer AL; ALLFTD consortium; Petrucelli L. Comprehensive cross-sectional and longitudinal analyses of plasma neurofilament light across FTD spectrum disorders. Cell Rep Med. 2022 Apr 19;3(4):100607. doi: 10.1016/j.xcrm.2022.100607. eCollection 2022 Apr 19. PMID 35492244
- See also: ALLFTD is the parent study of the NSP. — https://www.allftd.org/